CLINICAL TRIAL: NCT06658054
Title: Analgesic Efficacy of Erector Spinae Plane Block with Dexmedetomidine and Dexamethasone As Adjuvants in Single to Three-Level Lumbar Spine Fusion
Brief Title: Erector Spinae Plan Block (ESPB) with Dexmedetomidine and Dexamethasone in Lumbar Spine Fusion
Acronym: ESPB
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Paul S. Lee, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-23-00440
Record Dates: First submitted 2024-10-22; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Lumbar Degenerative Disease
Keywords: analgesia; ESPB; erector spinae plane block; dexmedetomidine; dexamethasone; bupivacaine; randomized; blinded; postoperative; opioid; PONV; nausea; vomitting; fusion
MeSH Terms: conditions — Agnosia; Postoperative Nausea and Vomiting; Nausea

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Spine Surgeon
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (control) (Active Comparator): Patients will receive an erector spinae plane block (ESPB) with 20 cc solution per single-shot injection comprised of 0.25% bupivacaine and 0.9% normal saline under ultrasound guidance to be administered bilaterally (40 cc total).
  Interventions: Drug: Control (Standard treatment)
- Group B (Intervention) (Active Comparator): Patients will receive ESPB with 20cc solution per single-shot injection comprised of 0.25% bupivacaine, 25mcg dexmedetomidine, and 5mg dexamethasone under ultrasound guidance to be administered bilaterally (40 cc total). This is in addition to the bupivacaine.
  Interventions: Drug: Adjuvant analgesia

INTERVENTIONS:
Drug: Adjuvant analgesia — Patients will receive adjuvant dexmedetomidine (25mcg) and dexamethasone (5mg) in addition to bupivacaine.
  Arms: Group B (Intervention)
Drug: Control (Standard treatment) — Patient will receive standard ESPB with bupivacaine and normal saline
  Arms: Group A (control)

SUMMARY:
This study wants to understand if using a pre-operative anesthetic injection could contribute to better pain relief after the surgery. This injection is referred to as an erector spinae plane block (ESPB, or "Block" for short). In the past, blocks have been commonly used to alleviate different types of pain, including pain following lumbar spine surgery, but our investigators are curious to study if adding two additional commonly used drugs could improve pain relief following surgery when used together. This possibility for improvement in pain management is important for our doctors to study because they want to find ways to reduce the amount of pain medication required after surgery.

We try to assess if one treatment is better than the other by looking into the amount of pain medication used immediately after the surgery (up to five times within the first 2 days; this is usually done by reviewing progress notes) and by asking patients if they can share with us their pain experienced at different times during their stay at the hospital and at 2-weeks after their procedure.

DETAILED DESCRIPTION:
Regional anesthetic techniques, including interfascial plane blocks, have demonstrated success in postoperative pain control and improved patient satisfaction. Erector spinae plane blocks (ESPB) are a relatively new regional anesthetic modality, which have shown potential for perioperative pain control in lumbar spinal surgery. This study aims to investigate whether adding dexmedetomidine and dexamethasone as adjuncts to bupivacaine in ESPB improves analgesia and reduces opioid usage in lumbar spinal fusion patients receiving multimodal pain regimens. It will also assess the impact of these adjuncts on postoperative nausea and vomiting (PONV) and anti-emetic medication requirements. The study employs a randomized, double-blind design, with participants divided into two groups: ESPB without adjuvants (Group A) and ESPB with dexmedetomidine and dexamethasone (Group B). Primary outcomes include opioid consumption at 24 hours postoperatively, while secondary outcomes involve opioid consumption at various time points and visual analog scale (VAS) pain scores. The results of this investigation will provide valuable insights into the efficacy of ESPB with adjuncts in postoperative pain management in lumbar spinal fusion patients.

ELIGIBILITY:
Inclusion Criteria:

* Medically optimized patients undergoing 1-3 level lumbar fusion surgery for treatment of degenerative lumbar spinal pathologies
* Aged 18 years or older
* English-speaking patients

Exclusion Criteria:

* Patients with surgical indications for infection, malignancy, or trauma
* women who are pregnancy or breastfeeding
* Patients with respiratory compromise
* Patients who are smokers
* Patients with allergies to local anesthetics, and/or opioid medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Postoperative opioid consumption | 24 hours postoperatively
  measured in morphine milligram equivalents (MME)

IPD SHARING:
Plan to Share IPD: Undecided
Aggregated data will be shared during publication.